CLINICAL TRIAL: NCT03291366
Title: Intrathecal Injection of Mesenchymal Stem Cells in Central Nervous System injury2017
Brief Title: Mesenchymal Stem Cells in Central Nervous System injury2017
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Principal Investigator, Jianming Tan, Professor, Fuzhou General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC-CNS2017
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Central Nervous System Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSC (Experimental): infusion of aUCMSC and conventional therapy
  Interventions: Drug: UCMSCC; Drug: conventional treatment
- conventional (Active Comparator): conventional therapy
  Interventions: Drug: conventional treatment

INTERVENTIONS:
Drug: UCMSCC — infusion of aUCMSC and conventional therapy
  Arms: MSC
Drug: conventional treatment — conventional treatment

SUMMARY:
Central nervous system (CNS) injury leads to morbidity in patients, which has few good rehabilitation measures. Mesenchymal stem cells seem to have regenerative and tissue-repairing capabilities. The investigators design this study to infuse mesenchymal stem cells (MSCs) intrathecally to CNS injury patients, and observe the safety and efficacy by recording the change of nervous system scores, trying to prove the effect of MSC in rehabilitate CNS injury.

ELIGIBILITY:
Inclusion Criteria:

* CNS injury > 3 months
* age > 18 years
* willing to give consent
* stable vital signs
* absence of active infectcion

Exclusion Criteria:

* any contradiction to intrathecal infusion
* age < 18 years
* CNS injury < 3 months
* CNS injury > 3 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
life quality score | 1y

SECONDARY OUTCOMES:
adverse events | 1y

IPD SHARING:
Plan to Share IPD: No